CLINICAL TRIAL: NCT06758687
Title: The Effect of Kinesio Taping Applied to Operating Room Nurses on Low Back Pain, Fatigue, and Sleep Quality: A Randomized Controlled Trial
Brief Title: The Effect of Kinesio Taping Applied to Operating Room Nurses on Low Back Pain, Fatigue, and Sleep Quality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Kezban KORAŞ, Assoc. Prof., Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Kinezyo2024
Record Dates: First submitted 2024-12-19; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Lower Back Pain; Kinesio Taping
Keywords: Operating room nurse; lower back pain; sleep quality; fatigue; kinesio taping
MeSH Terms: conditions — Low Back Pain; Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Introductory Information Form (No Intervention): It is a form prepared by the researcher in line with the literature, including questions such as age, professional experience, number of weekly working days, average daily surgery duration, exercise habits, smoking and alcohol consumption habits, musculoskeletal system problems, operating room conditions and equipment satisfaction.
- Visual Analog Skala (Experimental): VAS is used by having the patient mark the intensity of their pain on a 10 cm ruler ranging from "No pain" to "Unbearable pain".
  Interventions: Other: Kinesiotape Application
- Quebec Low Back Pain Disability Scale (Experimental): Includes a 20-item questionnaire to measure disability experienced during daily life activities. The five-point Likert-type scoring system used in this scale shows that the level of disability is high as the score increases
  Interventions: Other: Kinesiotape Application
- Visual Similarity Scale for Fatigue (Experimental): The 18-item scale developed by Yurtsever and Beduk in 2003, includes two subscales: fatigue and energy. While the items related to fatigue cover the items from 1 to 5 and 11 to 18, the items related to energy are from 6 to 10. Each item is evaluated on a 10 cm long line, from the most positive to the most negative expression or vice versa. High scores on the fatigue subscale and low scores on the energy subscale indicate increased fatigue.
  Interventions: Other: Kinesiotape Application
- Richard-Campbell Sleep Scale (Experimental): This scale evaluates six different factors such as the depth of night sleep, time it takes to fall asleep, frequency of awakenings, time it takes to stay awake, general quality of sleep, and environmental noise level. Each factor is scored between 0 and 100 using a visual analog scale. Scores between "0 and 25" indicate poor sleep quality, while scores between "76 and 100" indicate good sleep quality.
  Interventions: Other: Kinesiotape Application

INTERVENTIONS:
Other: Kinesiotape Application — Before the appropriate taping is applied to the waist area, a small piece of kinesio tape will be attached to the participant's thigh area and an allergy test will be performed. If the participant does not have any complaints within 5-10 minutes, the participant will be taped. The tape to be used in this study will be waterproof, porous, breathable, 5 cm wide and 0.5 mm thick.
  After the initial evaluation is completed, kinesio taping will be applied to the paravertebral muscles. First, the participant will be asked to perform trunk flexion while standing with their forearms supported by a table. While the participant is in this position, two "I" shaped tapes will be attached to the right and left sides of the spine (in the cranial direction) along the paravertebral muscle line without applying tension. Then, the field correction technique will be applied. While the participant is standing with their forearms supported on the table, four "I" tapes overlapping in
  Arms: Quebec Low Back Pain Disability Scale; Richard-Campbell Sleep Scale; Visual Analog Skala; Visual Similarity Scale for Fatigue

SUMMARY:
This study aims to determine the effects of kinesiology taping applied to operating room nurses on lower back pain, fatigue, and sleep quality. The research will be conducted using a randomized controlled experimental design with pre-test and post-test control groups. The universe of the study will consist of 100 operating room nurses working in a university hospital. The sample size has been calculated as a total of 84 nurses (Intervention group: 42; Control group: 42) based on power analysis calculations. The study will commence after obtaining the necessary permissions. Data collection will involve the use of the Descriptive Information Form, Visual Analog Scale, Quebec Back Pain Disability Scale, Visual Analogue Scale for Fatigue, and the Richards-Campbell Sleep Questionnaire. Participants who consent to the study will be administered the Descriptive Information Form, Visual Analog Scale, Quebec Back Pain Disability Scale, Visual Analogue Scale for Fatigue, and Richards-Campbell Sleep Questionnaire before the application of kinesiology tape. Subsequently, a physiotherapist from the research team will apply kinesiology tape to the paravertebral muscles using the muscle technique. As the literature suggests that the most suitable number of days for kinesiology tape application is four, participants will be instructed not to remove the tapes for four days. Additionally, participants will be informed that they can continue their daily activities and shower with the kinesiology tape on. The Visual Analog Scale will be applied to the participants at the end of the workday on the day of the kinesiology tape application and at the end of the workday for four days. At the end of the fourth day, all data collection tools will be applied. Seven days after the application, the scales will be filled out again by the nurses to determine if the effects of the kinesiology tape persist. Participants in the control group who agree to participate in the study will have data collected at the same time intervals as the intervention group participants using the same data collection tools. The Visual Analogue Scale will be administered to participants at the end of the day the data collection tools are filled out and at the end of the workday for four consecutive days. At the end of the fourth day, all data collection tools will be applied again. Seven days after the application, all scales will be refilled by the nurses..

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Working in the operating room for at least one year

Exclusion Criteria:

* Presence of conditions that will prevent the application of kinesio tape (excessive hair in the area where it is applied, skin rash, urticaria, etc.)
* Necessity for continuous use of analgesics

Exclusion Criteria for the Study

* Desire to leave the study while the study is ongoing
* Allergic reaction or skin irritation to kinesio tape during the study
* Use of analgesics during the period when kinesio tape is applied

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Skala | Before kinesio tape application
  VAS is used by having the patient mark the intensity of their pain on a 10 cm ruler ranging from "No pain" to "Unbearable pain".
Visual Analog Skala | 12 hours after kinesio tape application
  VAS is used by having the patient mark the intensity of their pain on a 10 cm ruler ranging from "No pain" to "Unbearable pain".
Visual Analog Skala | Kinesiotape application will be applied on the 2nd, 3rd and 4th days after work at 20:00 pm.
  VAS is used by having the patient mark the intensity of their pain on a 10 cm ruler ranging from "No pain" to "Unbearable pain".
Visual Analog Skala | Will be re-evaluated 7 days after the 4-day application (11th day)
  VAS is used by having the patient mark the intensity of their pain on a 10 cm ruler ranging from "No pain" to "Unbearable pain".
Quebec Low Back Pain Disability Scale | Before kinesio tape application
  Includes a 20-item questionnaire to measure disability experienced during daily life activities. The five-point Likert-type scoring system used in this scale shows that the level of disability is high as the score increases
Quebec Low Back Pain Disability Scale | 4th day of kinesio tape application at 08:00 pm
  Includes a 20-item questionnaire to measure disability experienced during daily life activities. The five-point Likert-type scoring system used in this scale shows that the level of disability is high as the score increases
Quebec Low Back Pain Disability Scale | Will be re-evaluated 7 days after the 4-day application (11th day)
  Includes a 20-item questionnaire to measure disability experienced during daily life activities. The five-point Likert-type scoring system used in this scale shows that the level of disability is high as the score increases
Visual Similarity Scale for Fatigue | Before kinesio tape application
  The 18-item scale developed by Yurtsever and Beduk in 2003, includes two subscales: fatigue and energy. While the items related to fatigue cover the items from 1 to 5 and 11 to 18, the items related to energy are from 6 to 10. Each item is evaluated on a 10 cm long line, from the most positive to the most negative expression or vice versa. High scores on the fatigue subscale and low scores on the energy subscale indicate increased fatigue.
Visual Similarity Scale for Fatigue | 4th day of kinesio tape application at 08:00 pm
  The 18-item scale developed by Yurtsever and Beduk in 2003, includes two subscales: fatigue and energy. While the items related to fatigue cover the items from 1 to 5 and 11 to 18, the items related to energy are from 6 to 10. Each item is evaluated on a 10 cm long line, from the most positive to the most negative expression or vice versa. High scores on the fatigue subscale and low scores on the energy subscale indicate increased fatigue.
Visual Similarity Scale for Fatigue | Will be re-evaluated 7 days after the 4-day application (11th day)
  The 18-item scale developed by Yurtsever and Beduk in 2003, includes two subscales: fatigue and energy. While the items related to fatigue cover the items from 1 to 5 and 11 to 18, the items related to energy are from 6 to 10. Each item is evaluated on a 10 cm long line, from the most positive to the most negative expression or vice versa. High scores on the fatigue subscale and low scores on the energy subscale indicate increased fatigue.
Richard-Campbell Sleep Scale | Before kinesio tape application
  This scale evaluates six different factors such as the depth of night sleep, time it takes to fall asleep, frequency of awakenings, time it takes to stay awake, general quality of sleep, and environmental noise level. Each factor is scored between 0 and 100 using a visual analog scale. Scores between "0 and 25" indicate poor sleep quality, while scores between "76 and 100" indicate good sleep quality.
Richard-Campbell Sleep Scale | 4th day of kinesio tape application at 08:00 pm
  This scale evaluates six different factors such as the depth of night sleep, time it takes to fall asleep, frequency of awakenings, time it takes to stay awake, general quality of sleep, and environmental noise level. Each factor is scored between 0 and 100 using a visual analog scale. Scores between "0 and 25" indicate poor sleep quality, while scores between "76 and 100" indicate good sleep quality.
Richard-Campbell Sleep Scale | Will be re-evaluated 7 days after the 4-day application (11th day)
  This scale evaluates six different factors such as the depth of night sleep, time it takes to fall asleep, frequency of awakenings, time it takes to stay awake, general quality of sleep, and environmental noise level. Each factor is scored between 0 and 100 using a visual analog scale. Scores between "0 and 25" indicate poor sleep quality, while scores between "76 and 100" indicate good sleep quality.

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study are not publicly available due protection of personal data of participants but are available from the corresponding author on reasonable request.